CLINICAL TRIAL: NCT01934543
Title: Differential Effects of Saturated and Polyunsaturated Fatty Acids on Chylomicron Secretion and Expression of Key Genes and Proteins That Regulate Intestinal Lipid Metabolism in Men With Dyslipidemia Associated With Insulin-resistance
Brief Title: Effects of Polyunsaturated Fatty Acids on Intestinal Lipid Metabolism in Insulin-resistant Men
Acronym: PUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-PUFA
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyunsaturated fatty acids diet (Experimental): During 4 weeks, subjects eat a diet high in polyunsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 6.0% from saturated fat; 14.4% from monounsaturated fat; 12.6% from n-6 polyunsaturated fat).
  Interventions: Other: Polyunsaturated fatty acids diet
- Saturated fatty acids diet (Experimental): During 4 weeks, subjects eat a diet high in polyunsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 13.4% from saturated fat; 15.3% from monounsaturated fat; 4.0% from n-6 polyunsaturated fat).
  Interventions: Other: Saturated fatty acids diet

INTERVENTIONS:
Other: Polyunsaturated fatty acids diet — During 4 weeks, subjects eat a diet high in polyunsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 6.0% from saturated fat; 14.4% from monounsaturated fat; 12.6% from n-6 polyunsaturated fat).
  Arms: Polyunsaturated fatty acids diet
Other: Saturated fatty acids diet — During 4 weeks, subjects eat a diet high in polyunsaturated fatty acids (percent of total caloric intake: 15.0% from proteins; 50.0% from carbohydrates; 35.0% from fat: 13.4% from saturated fat; 15.3% from monounsaturated fat; 4.0% from n-6 polyunsaturated fat).
  Arms: Saturated fatty acids diet

SUMMARY:
The overaccumulation of apolipoprotein (apo)B-48-containing lipoproteins of intestinal origin observed in patients with insulin-resistance is now thought to be attributable to both elevated intestinal production and reduced clearance of these lipoproteins. Substantial evidence exists indicating that elevated plasma levels of these lipoproteins are associated with increased cardiovascular disease (CVD) risk. Therefore, reduction of atherogenic plasma TRL levels of intestinal origin appears to be crucial to improve CVD risk associated with insulin-resistance. In this regard, there is some evidence that the clinical recommendation to replace dietary saturated fatty acids (SFAs) by n-6 polyunsaturated fatty acids (PUFAs) reduces CVD risk in the general population. Although the beneficial impact of n-6 PUFAs on CVD risk has been related primarily to favorable changes in plasma LDL-cholesterol levels, recent data suggest that chronic n-6 PUFA consumption may also exert beneficial effects on CVD risk by reducing postprandial lipemia. The impact of substituting SFAs by n-6 PUFAs on postprandial lipid response may be of even greater significance in dyslipidemic patients with insulin-resistance among whom intestinal triglyceride-rich lipoproteins (TRLs) represent a large proportion of the atherogenic lipoproteins. The general objective of the proposed research is to investigate how dietary n-6 PUFAs in place of SFAs modify intestinal lipoprotein metabolism in men with dyslipidemia associated with insulin-resistance. The investigators hypothesize that the intestinal secretion of apoB-48-containing lipoproteins will be lower following a diet rich in n-6 PUFAs than after consuming a diet rich in SFAs. The investigators also hypothesize that substitution of SFAs by n-6 PUFAs will be associated with significant alterations in expression of key genes and proteins involved in intestinal lipoprotein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18-60 years
* Waist circumference > 102 cm
* HDL-cholesterol < 1.1 mmol/L
* Triglycerides > 1.7 mmol/L
* Fasting blood glucose > 6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Women
* Men < 18 or > 60 years
* Smokers (> 1 cigarette/day)
* Body weight variation > 10% during the last 6 months prior to the study baseline
* Subjects with a previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with a monogenic dyslipidemia
* Subjects on hypertension medications or medications known to affect lipoprotein metabolism or the integrity of gastrointestinal mucosa
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in TRL apolipoprotein B48 (apoB-48) production rate. | At week 4 and week 12 (at the end of the two 4-weeks diets).

SECONDARY OUTCOMES:
Changes in duodenal expression of genes that regulate intestinal lipid absorption. | At week 4 and week 12 (at the end of the two 4-weeks diets).
  Genes that regulate intestinal lipid absorption that will be measured are Niemann-Pick C1-like 1 (NPC1L1), Adenosine triphosphate(ATP)-binding cassette transporters (ABCG5/8), Fatty Acid Binding Protein (FABP), Sterol Regulatory Element Binding Protein (SREBP-1c).
Changes in duodenal expression of genes that regulate intestinal lipid synthesis. | At week 4 and week 12 (at the end of the two 4-weeks diets).
  Genes that regulate intestinal lipid synthesis that will be measured are Acyl-Coenzyme A(CoA):diacylglycerol acyltransferase (DGAT), Acyl-CoA:cholesterol O-acyltransferase 2 (ACAT2) and 3-hydroxy-methylglutaryl-CoA reductase (HMG CoA reductase).
Change in synthesis of apoB-48 containing lipoproteins (Microsomal triglyceride transfer protein (MTP), apoB-48). | At week 4 and week 12 (at the end of the two 4-weeks diets).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD,FRCP,PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada

REFERENCES:
- [Derived] Drouin-Chartier JP, Tremblay AJ, Lepine MC, Lemelin V, Lamarche B, Couture P. Substitution of dietary omega-6 polyunsaturated fatty acids for saturated fatty acids decreases LDL apolipoprotein B-100 production rate in men with dyslipidemia associated with insulin resistance: a randomized controlled trial. Am J Clin Nutr. 2018 Jan 1;107(1):26-34. doi: 10.1093/ajcn/nqx013. PMID 29381796